CLINICAL TRIAL: NCT00114621
Title: Anthrax Vaccine Clinical Trials
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040283; 04-CH-0283
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-16

CONDITIONS: Anthrax
Keywords: PA; Phase I; Phase 2; Safety; Immunogenicity
MeSH Terms: conditions — Anthrax | interventions — Anthrax Vaccines; Blood Chemical Analysis; Hematologic Tests; Urinalysis

INTERVENTIONS:
Drug: Anthrax Vaccine
Procedure: Blood Chemistry
Procedure: Hematology
Procedure: Urinalysis

SUMMARY:
This study will examine the recombinant, that is, produced by genetic engineering, protective antigen (rPA) that brings about antibodies to neutralize the anthrax toxin and that could therefore be predicted to offer protection against anthrax. Today, anthrax is rarely encountered in the United States, since the introduction of vaccines for cattle in the 1930s. A human vaccine was licensed in 1970. Vaccination against anthrax has been confined to people at risk, such as wool sorters and some veterinarians. However, the rising prospects of B. anthracis being used as a weapon have led to routine administration of the anthrax vaccine to members of the armed forces.

Adults who are in good health may be eligible for this study. The involvement of 300 adults is planned.

Participants will have a general physical exam and test for vital signs. There will also be collection of blood for chemistry and hematology; urinalysis; tests for HIV, hepatitis B and C, and liver function; and a pregnancy test, if applicable.

On a random basis, patients will receive one of the rPA formulations. Two doses of rPA will be evaluated, 10 microgram ((Micro)g) and 20 (Micro)g. This evaluation aims to establish the safety and most desirable level of dosage. Patients will receive one injection of the vaccine, administered in the left shoulder or left thigh. About 30 minutes later, their temperature will be taken, and the injection site will be inspected. Rare but severe reactions could occur if there is extreme sensitivity to a vaccine. However, such an occurrence is extremely rare following a vaccine, and if there are any dangerous symptoms, they can be effectively treated by medications available to patients while they are at the clinic. If there are no significant abnormal results, patients may return home. About 6 hours later and daily for 7 days, they will take their temperature and examine the injection site. The vaccine may cause temporary discomfort at the site of injection, and participants may experience a mild fever for 1 or 2 days after vaccination.

Patients will receive diary cards, a digital thermometer, and instructions on taking their temperature and measuring redness and swelling at the injection site, as well as for recording aches, muscle pain, or sensitivity to light for 7 days. They will be examined at the clinic at 72 hours following vaccination and also on the 7th day if they have a fever at or above 100.4 , if swelling is at or more than 2 inches, or if they request an exam. Meanwhile, a clinic staff member will call patients and discuss the findings. Then patients will receive a second and third injection of the same vaccine at 2-month intervals. There will also be interviews about patients' health at each visit to the clinic, plus monitoring of the vaccination after 6 hours and for 7 days. One year later, patients will receive a fourth injection of the same vaccine.

Direct benefit to participants in this study is not guaranteed, although an antibody response is predicted. The results in this study will help in the development of improved vaccines for anthrax.

DETAILED DESCRIPTION:
Anthrax is rarely encountered in the U.S. since the introduction of attenuated vaccines for cattle in the 1930's. A vaccine for humans, composed of a cell-free preparation absorbed onto alum, was licensed in 1970 after successful clinical trials. Vaccination against anthrax in the U.S. was confined to individuals at risk such as wool sorters and some veterinarians until the prospects were raised of B. anthracis being used as a weapon after the Iraq war. Now anthrax vaccine is administered routinely to the armed forces. Interest in improving this vaccine was stimulated by the use of B. anthracis spores for bioterrorism.

The active component of the investigational vaccine is called the protective antigen. When B. anthracis invades the host tissues, the protective antigen activates two other proteins to form anthrax toxin. The symptoms of anthrax are caused by this toxin. Alone, the protective antigen has no known toxicity. The gene for this protein has been isolated and changed specifically to improve its properties as a vaccine-this recombinant protective antigen (rPA) elicits antibodies that neutralize the anthrax toxin and, thereby, can be predicted to confer protection.

This is the first study of our investigational rPA vaccine in humans. The broad objectives are to characterize the safety and serum antibody levels of different doses and formulations of rPA in comparison to the licensed anthrax vaccine, AVA.

ELIGIBILITY:
* INCLUSION CRITERIA: Phase I

Healthy 18 to 45 year-olds of either sex.

EXCLUSION CRITERIA:

Patients receiving chronic medication, are pregnant or intend to become pregnant during the study.

Individuals who are HIV positive, have abnormal liver function, had anthrax, or received anthrax vaccine, have received or intend to receive an experimental vaccine or medication within 30 days of injection of the experimental anthrax vaccine.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2004-09-08; Study Completion 2011-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay W. Mash, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - Georgetown University, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] KEPPIE J, HARRIS-SMITH PW, SMITH H. THE CHEMICAL BASIS OF THE VIRULENCE OF BACILLUS ANTHRACIS. IX. ITS AGGRESSINS AND THEIR MODE OF ACTION. Br J Exp Pathol. 1963 Aug;44(4):446-53. No abstract available. PMID 14079018
- [Background] Turnbull PC, Leppla SH, Broster MG, Quinn CP, Melling J. Antibodies to anthrax toxin in humans and guinea pigs and their relevance to protective immunity. Med Microbiol Immunol. 1988;177(5):293-303. doi: 10.1007/BF00189414. PMID 3139974
- [Background] Schneerson R, Robbins JB, Taranger J, Lagergard T, Trollfors B. A toxoid vaccine for pertussis as well as diphtheria? Lessons to be relearned. Lancet. 1996 Nov 9;348(9037):1289-92. doi: 10.1016/S0140-6736(96)05243-9. No abstract available. PMID 8909384